CLINICAL TRIAL: NCT06681675
Title: The Effect of the Intrapartum Care Model Given in Line With WHO Recommendations on Labor Pain, Fear, Comfort, Duration, Oxytocin Use and Midwifery Care Perception: A Randomized Controlled Trial
Brief Title: The Effect of the Intrapartum Care Model Given in Line With WHO Recommendations on the Birth Process and Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Associate Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/671
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Birth Outcomes; Labor Pain and to Reduce Pain; Fear of Birth; Birth Comfort; Perception of Midwifery Care; Birth Period; Oxytocin Deficiency; WHO Intrapartum Care Recommendations
Keywords: WHO intrapartum care recommendations; Labor pain and to reduce pain; fear of birth; birth comfort; perception of midwifery care; Birth period; Oxytocin Deficiency
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (No Intervention): No intervention was made to the primiparous pregnant women in the control group other than routine intrapartum care applied in the hospital. After being admitted to the hospital for delivery, the pregnant women in the control group were informed about the study. Written consent was obtained. A personal information form was applied at the first clinic admission. When the cervical dilatation was 5 cm, VAS, Fear of Childbirth and Childbirth Comfort scales were applied. When the cervical dilatation was 9 cm, the labor monitoring form, VAS, Fear of Childbirth and Childbirth Comfort scales were applied. The routine practices and care of the maternity ward affiliated to the hospital were performed (anamnesis was taken, file was filled, intravenous access was established, routine blood tests were taken, vital signs were taken, enema was performed, vaginal examination every two hours and cervical changes were recorded on the partograph, continuous EFM (Electronic Fetal Monitoring) was applied
- The group that applied the Intrapartum Care Model (Experimental): In pregnant women with cervical dilatation of 5 cm, the Personal Information Form was completed at the initial clinic admission. •The Intrapartum Care Model was implemented for all primiparous pregnant women assigned to the intervention group during labor and after delivery by the researcher midwife, in accordance with the World Health Organization's positive birth recommendations. Data were collected using the Personal Information Form, Labor and Postpartum Follow-up Form, Visual Analog Scale (VAS), Labor Comfort Scale (CSC), Intrapartum Fear of Labor Scale, and Women's Perception of Supportive Care Given During Labor Scale. VAS, CSC, and Fear of Labor Scale were applied to women when cervical dilation was 5 cm and 9 cm. After delivery, the Women's Perception of Supportive Care Given During Labor Scale was applied.
  Interventions: Procedure: The group that applied the Intrapartum Care Model

INTERVENTIONS:
Procedure: The group that applied the Intrapartum Care Model — In pregnant women with cervical dilatation of 5 cm, the Personal Information Form was completed at the initial clinic admission.
  •The Intrapartum Care Model was implemented for all primiparous pregnant women assigned to the intervention group during labor and after delivery by the researcher midwife, in accordance with the World Health Organization's positive birth recommendations.
  Data were collected using the Personal Information Form, Labor and Postpartum Follow-up Form, Visual Analog Scale (VAS), Labor Comfort Scale (CSC), Intrapartum Fear of Labor Scale, and Women's Perception of Supportive Care Given During Labor Scale. VAS, CSC, and Fear of Labor Scale were applied to women when cervical dilation was 5 cm and 9 cm. After delivery, the Women's Perception of Supportive Care Given During Labor Scale was applied.
  Arms: The group that applied the Intrapartum Care Model

SUMMARY:
This study aimed to evaluate the effects of the intrapartum care model provided in line with the World Health Organization (WHO) recommendations on labor pain, fear, comfort, duration, oxytocin use and perception of midwifery care.

DETAILED DESCRIPTION:
The research is a randomized controlled trial. The research was conducted with 124 primiparous pregnant women (intervention group n=62, control group n=62) who were hospitalized in the delivery unit of Aksaray Training and Research Hospital between September 2023 and January 2024. The pregnant women in the intervention group were given the intrapartum care model in line with WHO recommendations after cervical dilation reached 5 cm. The control group received only the standard intrapartum care in the hospital. Data were collected using the personal information form, labor and postpartum follow-up form, Visual Analog Scale (VAS), Labor Comfort Scale (DKS), Intrapartum Fear of Labor Scale, and Women's Perception of Supportive Care Given During Childbirth Scale. VAS, DKS, and Fear of Childbirth scale were applied to women in both groups when cervical dilation was 5 cm and 9 cm. After birth, the Women's Perception of Supportive Care Given During Childbirth scale was applied.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* History of term pregnancy (38-42 weeks),
* Having a primiparous,
* Single, healthy, vertex positioned fetus,
* Having no complications that may cause dystocia in labor (such as contraction anomalies, birth object,
* Birth canal dystocia, dystocia related to the mother's psychology),
* Having a partner/husband,
* History of cervical dilatation of 5 cm or more,
* Being able to speak and understand Turkish

Exclusion Criteria:

* Those with maternal and fetal complications (oligohydramnios and polyhydramnios, placenta previa, preeclampsia, premature membrane rupture, presentation anomalies, intrauterine growth retardation, fetal anomalies, intrauterine death, macrosomic baby, etc.),
* Those with any complications that prevent vaginal delivery,
* Elective caesarean section, those who became pregnant with assisted reproductive techniques,
* Those who are multiparous,
* Those who have chronic diseases (such as hypertension, diabetes, heart disease).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Comparison of pre-intervention sociodemographic of pregnant women | 6 months
  Sociodemographic of pregnant women will be collected through surveys and compared and reported
Comparison of pre-intervention obstetric features of pregnant women | 6 months
  Obstetric of pregnant women will be collected through surveys and compared and reported.
Comparison of labor characteristics of pregnant women before intervention | 6 months
  Labor Characteristics of pregnant women will be collected through questionnaires and compared and reported.
Comparison of postpartum characteristics of pregnant women | 6 months
  Postpartum characteristics of pregnant women will be collected through surveys and compared and reported.
Comparison of duration of labor of groups | 6 months
  The duration of labor of the groups will be collected through surveys and compared and reported.
Comparison of pregnant women's VAS (pain perception) mean scores by groups | 6 months
  VAS (pain perception) scale will be applied to pregnant women. The pain scale (VAS) is 1-10 points (min-max), and as the score increases, women's pain perception also increases.
Comparison of pregnant women's fear of childbirth average scores by groups | 6 months
  A fear of childbirth scale will be applied to pregnant women. The fear of childbirth scale is 10-100 points (min-max), and as the score increases, women's fear of childbirth increases.
Comparison of pregnant women's birth comfort score averages by groups | 6 months
  A birth comfort scale will be applied to pregnant women. The birth comfort scale is 9-45 points (min-max), and as the score increases, women's birth comfort increases.
Comparison of mean scores of the scale of women's perception of supportive care given during childbirth by groups | 6 months
  A scale of women's perception of supportive care given during childbirth will be applied to pregnant women. The scale of women's perception of supportive care given during childbirth is 33-132 points (min-max), and as the score increases, women's perception of care increases.
Comparison of oxytocin use by groups | 6 months
  Oxytocin use by groups will be collected via survey and reported by comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan Çankaya, Assoc.Prof, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangir Meler K, Cankaya S. The effect of intrapartum care model given in line with World Health Organization (WHO) recommendations on labor pain, fear of labor, comfort of labor, duration of labor, administration of oxytocin and perception of midwifery care: a randomized controlled study. Postgrad Med. 2025 Jun;137(5):379-395. doi: 10.1080/00325481.2025.2501943. Epub 2025 May 11. PMID 40314363